CLINICAL TRIAL: NCT04816617
Title: A 12-month，Parallel-group, Randomised Controlled Exercise Trial in Young People With and Without Subthreshold Depression
Brief Title: The Effect of Exercise on Cognition and Preventing Depression in Young People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Psychiatric Hospital (Other Government)
Collaborators: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, Kangguang Lin, MD.PhD, Guangzhou Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Exercise, Cogntion and MDD
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Subthreshold Depression; Exercise; Clinically-well; Cognitive Change
Keywords: Subthreshold depression, aerobic exercise, Major depression, Intervention; Cognition
MeSH Terms: conditions — Motor Activity; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Experimental): The whole exercise lasts for 12 months, consisted of 6-month supervised exercise and 6-month maintenance period. It is moderate -intensity exercise (60-80% Maximum heart rate), each time last for 30 mins (plus 10-minutes for warm-up and cool-down), 3-4 times a week, for the first six months, which will be supervised in person by physical educators and/or physical professionals. In the maintenance period, participants are asked to exercise at the same intensity and frequency, but will not be supervised in person by physical educators/professionals. They will receive reminder on a weekly basis and their physical activities be recorded by accelerometer. Types of exercise will be chosen according to individual school's facility and feasibility, including jogging, fast walking, badminton, running, football etc.
  Interventions: Behavioral: Aerobic exercise intervention
- Psycho-education (Placebo Comparator): It consists of 6 sections of psycho-education, with topics covering mood regulations and mental well-being. Approximately 1 section in every two months.
  Interventions: Behavioral: Psycho-education

INTERVENTIONS:
Behavioral: Aerobic exercise intervention — The whole exercise lasts for 12 months, consisted of 6-month supervised exercise and 6-month maintenance period. It is moderate -intensity exercise (60-80% Maximum heart rate), each time last for 30 mins (plus 10-minutes for warm-up and cool-down), 3-4 times a week, for the first six months, which will be supervised in person by physical educators and/or physical professionals. In the maintenance period, participants are asked to exercise at the same intensity and frequency, but will not be supervised in person by physical educators/professionals. They will receive reminder on a weekly basis and their physical activities be recorded by accelerometer. Types of exercise will be chosen according to individual school's facility and feasibility, including jogging, fast walking, badminton, running, football etc.
  Arms: Aerobic Exercise
Behavioral: Psycho-education — It consists of 6 sections of psycho-education, with topics covering mood regulations and mental well-being. Approximately 1 section in every two months.
  Arms: Psycho-education

SUMMARY:
It is estimated that approximately 30% of child and adolescents manifest subthreshold depression (including other specified depressive disorder and unspecified depressive disorder), which can further develop into major depression with as high as 25%-50% within one year. The cognitive development of adolescents is a critical area of research, given its significant implications for academic performance, mental health, and overall well-being. During adolescence, the brain undergoes substantial structural and functional changes, particularly in regions associated with executive function, memory, and processing speed. These changes provide a unique opportunity to explore interventions that can support and enhance cognitive development. One such promising intervention is physical exercise. Adolescence is characterized by rapid cognitive growth, including improvements in executive functions such as planning, decision-making, and inhibitory control. These cognitive abilities are essential for academic success and social interactions. However, this period also presents risks for cognitive and emotional disturbances, making it vital to identify effective strategies to promote healthy cognitive development. Despite the promising evidence, there is a need for more rigorous research, particularly long-term randomized controlled trials (RCTs), to establish the causal relationship between exercise and cognitive function in adolescents, including those with sub-threshold depression. Most existing studies have focused on short-term interventions or specific cognitive tasks, leaving a gap in our understanding of the sustained effects of exercise over an extended period. Additionally, the transition from supervised to unsupervised exercise and its impact on adherence and cognitive outcomes is underexplored. There is also a need to evaluate the potential of exercise as a preventive strategy against the development of major depressive disorder in this vulnerable population. Additionally, evidence suggests that participants with lower baseline levels of physical activity may experience more significant cognitive improvements from exercise interventions than those with higher baseline activity levels. This highlights the importance of considering baseline physical activity levels when assessing the effectiveness of exercise on cognitive outcomes.

This study will particularly focus on the cognitive domains of attention, memory, and processing speed. These domains are critical for academic success and daily functioning and are often impacted in adolescents with sub-threshold depression. Previous research has shown that these domains are particularly responsive to physical exercise interventions.

DETAILED DESCRIPTION:
This is multi-center, psycho-education randomized controlled trial, consisting of two periods with each of 6 months (i.e supervised and maintenance period). In the exercise intervention arm, during the first 6 months, participants will be asked to do moderate-intensity aerobic exercise 3-4 times a week, which will be supervised in person by physical educators/professionals. In the next 6-month maintenance period, participants will be asked to continue doing aerobic exercise at the same intensity and frequency, which will not be supervised in person by educators/professionals, but they will be sent reminders and report adherence monthly. All of the physical activity will be recorded by accelerometer at scheduled time points (e.g. the first week, 6 week, 3 month, 6 month, 9 month, 12 month). Psycho-education group will be given 6 sections of general psycho-education onsite and/or virtually dependent on the surroundings with regards to the impact of the COVID-19 pandemic. The main aim of this trial is to investigate the effect of long-term aerobic exercise on cognition and prevention depression in young people with or without subthreshold depression.

ELIGIBILITY:
Inclusion Criteria:

* PHQ-9 ≥5
* 12~17 years old.

Exclusion Criteria:

* Current or past DSM-5 criteria for major depressive disorder,Bipolar disorder, Schizophrenia.
* Musculoskeletal problems such as arthritis, gout, osteoporosis, or back, hip or knee pain that may interfere with exercising
* A history of organic brain disease or brain trauma
* Alcohol, drug or other psychoactive substance abuse or dependence
* Currently enrolled in another exercise study
* Any conditions that would make exercise unsafe or unwise
* Taking medication that interferes with heart rate response to exercise such as beta blockers

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 628 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Attention measure by Choice Reaction Time task (CRT) incorporated into THINC-it® | month 12
  Attention will be measured by the Choice Reaction Time task (CRT).

SECONDARY OUTCOMES:
The rate of occurrence of MDD | Month 6 and month 12
  Kiddie-Sads-Present and Lifetime Version (K-SADS-PL)
Levels of inflammatory biomarkers from baseline | Month 6 and month 12
  inflammatory biomarkers (IL-6, CRP etc) will be analyzed using ELISA
Occurrence of Non-suicidal self-injury and suicidal behavior | Month 6 and month 12
Physical activity level | Month 6 and 12
  The International Physical Activity Questionnaire - Short Form (IPAQ - SF) will be used to assess physical activity level
P Wave changes over time | Month 6 and 12
  Brain activity will be detected by Electroencephalograph (EEG)
New onset of subthreshold depression in healthy volunteers | Month 6 and 12
  subthreshold depression is defined by DSM-5 Other specified Depressive Disorder and Unspecified Depressive Disorder
Changes from baseline in memory measured N-back memory task (N-BACK) | month 6 and month 12
  N-back memory task (N-BACK) was used to measure short-term memory.
Changes from baseline in subjective cognition measured by Perceived Deficits Questionnaire 5 (PDQ-5) | Month 6 and 12
  Perceived Deficits Questionnaire 5 (PDQ-5) is a subjective measure, which broadly evaluates attention/concentration, planning/organisation, as well as retrospective and prospective memory.
Changes from baseline in Processing Speed. | Month 6 and 12
  Digit Symbol Substitution Test (DSST) was used to measure Processing Speed.
Changes from baseline in executive function. | Month 6 and 12
  Trail Making Test-B (TMT-B) was used to measure Executive function.
Changes from baseline in Attention measure by Choice Reaction Time task (CRT) | month 6
  Attention measure by Choice Reaction Time task (CRT)

CONTACTS AND LOCATIONS:
Overall Officials: Kangguang Lin, MD,PhD, Study Director — The Affiliated Brain Hospital of Guangzhou Medical University; Tifei Yuan, PhD, Principal Investigator — Shanghai Mental Health Center; Kwok-Fai So, PhD, Study Chair — Jinan University
Locations (1):
- The first Huaiji middle school, Shaoxing, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Werneck AO, Tian X, Lu W, Li D, Liu T, Wu S, Li X, Wang R, Gao Y, Li X, Chen J, Vancampfort D, Solmi M, Fabiano N, Schuch F, Plener PL, McIntyre RS, So KF, Stubbs B, Lin K. Can exercise reduce the risk of suicidal ideation and behaviors in youth at school? A 12-month cluster randomized control trial. J Psychiatr Res. 2025 Dec 11;194:71-78. doi: 10.1016/j.jpsychires.2025.12.025. Online ahead of print. PMID 41448028